CLINICAL TRIAL: NCT07169994
Title: A Multi-center, Open-Label, Phase Ib/II Study of YL202 in Combination With Anti-tumor Therapy to Evaluate the Safety, Tolerability, and Efficacy in Patients With Advanced Solid Tumors
Brief Title: A Study of YL202 in Combination With Other Anti-tumor Therapies in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL202-CN-204-02
Record Dates: First submitted 2025-09-03; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors; Breast Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Injections; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YL202 in combination with Toripalimab (Experimental): Part 1 (dose escalation stage and backfill stage) & Part 3 (dose expansion stage): YL202 for injection in combination with Toripalimab injection
  Interventions: Drug: YL202 for injection; Toripalimab injection
- YL202 in combination with Furmonertinib Mesilate (Experimental): Part 2 (dose escalation stage and backfill stage) & Part 4 (dose expansion stage): YL202 for injection in combination with Furmonertinib Mesilate Tablets
  Interventions: Drug: YL202 for injection; Furmonertinib Mesilate Tablets

INTERVENTIONS:
Drug: YL202 for injection; Toripalimab injection — Part 1: YL202 and Toripalimab will be administered intravenously.
  Part 3: participants will receive escalating doses of YL202 and fixed dose of Toripalimab until YL202 doses for optimization are determined.
  Dose expansion stage: participants will receive a dose of YL202 not exceeding the maximum dose level achieved during the dose-escalation stage and fixed dose of Toripalimab
  Arms: YL202 in combination with Toripalimab
Drug: YL202 for injection; Furmonertinib Mesilate Tablets — Part 2: YL202 will be administered intravenously，Furmonertinib Mesilate Tablets will be administered orally.
  Dose escalation stage: participants will receive escalating doses of YL202 and fixed dose of Furmonertinib Mesilate until YL202 doses for optimization are determined.
  Part 4: participants will receive a dose of YL202 not exceeding the maximum dose level achieved during the dose-escalation stage and fixed dose of Furmonertinib Mesilate.
  Arms: YL202 in combination with Furmonertinib Mesilate

SUMMARY:
This is a multicenter, open-label, phase Ib/II study of YL202 in combination with other anti-tumor therapies to Evaluate the Safety, Tolerability, and Efficacy in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the study before the start of the study and voluntarily sign their name and date in the informed consent form (ICF)
2. Able and willing to comply with protocol visits and procedures
3. Aged between 18 to 75 years
4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
5. Previously treated by standard treatment or have not been treated for metastatic setting;
6. Adequate organ and bone marrow function.
7. Have at least 1 extracranial measurable tumor lesion.
8. Adequate archival formalin-fixed paraffin embedded （FFPE） tissue from prior biopsy.

Exclusion Criteria:

1. With prior drug therapy targeting HER3 (including antibodies, antibody-drug conjugates [ADCs]), chimeric antigen receptor T-cell immunotherapy (CAR-T), and other drugs).
2. Previously intolerant to topoisomerase I inhibitors or ADC therapy composed of topoisomerase I inhibitors.
3. Are participating in another clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study.
4. The washout period from the previous anti-tumor therapy is insufficient before the first dose of the investigational product.
5. Patients who have received major surgery (excluding diagnostic surgery) within 4 weeks before the first dose of the investigational product or those who are expected to receive major surgery during the study.
6. Prior treatment with allogeneic bone marrow transplantation or solid organ transplantation.
7. Prior treatment with systemic steroids (prednisone > 10 mg/day or equivalent) or other immunosuppressive treatment within 2 weeks before the first dose of the investigational product.
8. Patients who have received any live vaccine within 4 weeks before the first dose of the investigational product or those who plan to receive live vaccine during the study period.
9. With meningeal metastasis or cancerous meningitis.
10. With brain metastasis or spinal cord compression.
11. Patients with uncontrolled or clinically significant cardiovascular diseases.
12. Clinically significant complicated pulmonary disorders.
13. Patients diagnosed with Gilbert syndrome.
14. Those with uncontrolled effusion in the third space requiring repeated drainage.
15. With a medical history of gastrointestinal perforation and/or fistula within 6 months before the first dose, or with active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases that may lead to hemorrhage or perforation according to the investigator.
16. With serious infection before the first dose.
17. With known human immunodeficiency virus (HIV) infection.
18. With active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
19. With a medical history of any other primary malignancies within 5 years before the first dose of the investigational product.
20. Unrelieved toxicity of previous anti-tumor therapy.
21. With a history of severe hypersensitivity to inactive ingredients in the raw materials and drug product or other monoclonal antibodies.
22. Lactating women, or women who are confirmed pregnant via a pregnancy test within 3 days before the first dose.
23. With any diseases, medical conditions, organ system dysfunction, or social conditions that may interfere with the ability of subjects to sign the ICF, adversely affect the ability of subjects to cooperate and participate in the study, or affect the interpretation of study results, including but not limited to mental illness or substance/alcohol abuse, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Nature and frequency of dose-limiting toxicity (DLT) | 21 days after the first dose was administered to each subject.
  The purpose of DLT is to find maximum tolerated dose (MTD).
Nature and frequency of adverse events (AEs) | 42 days after the end of treatment (EOT).
  Nature and frequency of AEs with severity is aim to evaluate the safety of YL202 combination.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 3 years.
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Characterize Pharmacokinetics (PK) parameter AUC | Up to approximately 3 years
  The area under curve: AUC is the total amount of YL217 in bloodstream after drug administration.
Characterize Pharmacokinetics (PK) parameter Cmax | Up to approximately 3 years
  Maximum concentration: The highest measured concentration of YL217 in the bloodstream.
Characterize Pharmacokinetics (PK) parameter Ctrough | Up to approximately 3 years
  Trough concentration
Characterize Pharmacokinetics (PK) parameter Tmax | Up to approximately 3 years
  Time to maximum observed concentration
Characterize Pharmacokinetics (PK) parameter CL | Up to approximately 3 years
  Clearance： defined as the amount of drug removed from the bloodstream by the body per unit of time
Characterize Pharmacokinetics (PK) parameter Vd | Up to approximately 3 years
  volume of distribution
Characterize Pharmacokinetics (PK) parameter t1/2 | Up to approximately 3 years
  Half-life time：defined as the time it takes for the concentration of the drug in plasma or serum to be reduced by 50%
Immunogenicity endpoint: Incidence of anti-YL202 antibody (ADAs). | Up to approximately 3 years
  The presence of ADAs in patients treated with YL202 will be assessed to evaluate immunogenicity.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Anhui Provincial Hospital(The First Affiliated Hospital of Ustc), Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Meizhou People's Hospital（Huangtang Hospital）Meizhou Academy of Medical Sciences, Meizhou, Guangdong
  - Ghang xi Medical University Cancer Hospital, Nanning, Guangxi
  - Affiliated Hospital Of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Jiangsu Province Hospital（The First Affiliated Hospital With Nanjing Medical University, Jiangsu Women And Children Health Hospital), Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital Dalian University, Dalian, Liaoning
  - Liaoning cancer hospital &institute, Shenyang, Liaoning
  - Affiliated Zhongshan Hospital Dalian University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences&Sichuan Provincial People's Hospital, Sichuan, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality